CLINICAL TRIAL: NCT06549582
Title: Effect of Taohong Tongluo Xiaoban Prescription on Reprogramming of Lipid Metabolism and Endothelial Injury for Cerebral Infarction Patients：a Randomized Controlled Clinical Trial
Brief Title: Th Tl Xb Prescription on Reprogramming of Lipid Metabolism and Endothelial Injury for Cerebral Infarction Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yan Zhu (Other)
Responsible Party: Sponsor-Investigator, Yan Zhu, Principal Investigator, Beijing Electric Power Hospital
Organization: Beijing Electric Power Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Th Tl Xb PrescriptionlY2024007
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Infarction; Chinese Herbal Medicine; Clinical Trial; Lipid Metabolism Disorder; Endothelial Injury
MeSH Terms: conditions — Cerebral Infarction; Lipid Metabolism Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Fundamental medical treatment+Taohong Tongluo Xiaoban Prescription Incorporating the Taohong Tongluo Xiaoban prescription, which includes Pinelliae Rhizoma, Poria, Bambusae caulis in taenias, Aurantii Fructus Immaturus, Arisaema cum bile, Acori Tatarinowii Rhizoma, Persicae Semen, Carthami Flos, Chuanxiong Rhizoma and Paeoniae Radix Rubra as a once - daily dosage with one administration per dose.
  Interventions: Other: Taohong Tongluo Xiaoban Prescription; Other: Fundamental medical treatment
- control group (Active Comparator): Fundamental medical treatment The specific methods were developed in accordance with the 2010 Chinese Guidelines for Secondary Prevention of Ischemic Stroke and Transient Ischemic Attack. It primarily involves managing risk factors such as hypertension, diabetes, abnormal lipid metabolism, etc., and implementing antithrombotic therapy including antiplatelet agents (aspirin, clopidogrel, dipyridamole, dipyridamole + aspirin, clopidogrel + aspirin, silostazole, triflurosal, etc). For the management of post-stroke mood disorders, cognitive impairments, and spastic paralysis, pharmacological interventions encompass oral administration of anxiolytic or antidepressant agents, anti-dementia medications, as well as muscle relaxants.
  Interventions: Other: Fundamental medical treatment

INTERVENTIONS:
Other: Taohong Tongluo Xiaoban Prescription — Chinese herbal medicine "Taohong Tongluo Xiaoban prescription", which includes Pinelliae Rhizoma, Poria, Bambusae caulis in taenias, Aurantii Fructus Immaturus, Arisaema cum bile, Acori Tatarinowii Rhizoma, Persicae Semen, Carthami Flos, Chuanxiong Rhizoma and Paeoniae Radix Rubra as a once - daily dosage with one administration per dose
  Arms: intervention group
Other: Fundamental medical treatment — The specific methods were developed in accordance with the 2010 Chinese Guidelines for Secondary Prevention of Ischemic Stroke and Transient Ischemic Attack. It primarily involves managing risk factors such as hypertension, diabetes, abnormal lipid metabolism, etc., and implementing antithrombotic therapy including antiplatelet agents (aspirin, clopidogrel, dipyridamole, dipyridamole + aspirin, clopidogrel + aspirin, silostazole, triflurosal, etc). For the management of post-stroke mood disorders, cognitive impairments, and spastic paralysis, pharmacological interventions encompass oral administration of anxiolytic or antidepressant agents, anti-dementia medications, as well as muscle relaxants.

SUMMARY:
This study is a prospective, open-label, randomized control trial. It is planning to include 160 cerebral infarction patients which will be randomized in a 1﹕1 fashion to receive Chinese herbal medicines combined basic medicine treatment, or to receive standard basic medicine treatment within 3 months after inclusion. Follow-up will be performed after the treatment for 3 months to evaluate the incidence and disability rates of limb impairment, language impairment, cognitive impairment, and emotional disorders. The primary outcome is modified Rankin Scale Score, which is measured by the overall distribution from 0 (no symptoms) to 6 (death). The secondary outcome include the Evaluation of Neurological Function Deficit score (National Institute of Health stroke scale scoring) and carotid atherosclerotic plaque score (Crouse scoring system for neck carotid atherosclerotic plaque scoring). Additional outcomes include laboratory indicator to analysis the reprogramming of lipid metabolism and endothelial Injury, Chinese medicine symptom and sign scoring system and biological indicators. The investigators will perform the intention-to-treat analysis for withdrawal and missing data, and estimate the health economic value.

ELIGIBILITY:
Inclusion Criteria:

1. The CT/MRI examination findings were consistent with the diagnosis of Western cerebral infarction, aligning with the TCM apoplexy diagnosis. Primary stroke occurred 35±5 days ago.
2. The National Institutes of Health Stroke Scale (NIHSS) evaluates a range of scores from 4 to 24.
3. Coronary atherosclerotic heart disease is confirmed through coronary CT angiography. Carotid artery ultrasonography is employed to ascertain the presence or absence of plaque formation, with stable plaques exhibiting predominantly high and uneven echogenicity, while unstable plaques displayed low echo or irregular hypoechoic regions.
4. Age range: ≥35 years to ≤80 years.
5. First onset requires; patients with previous diseases and no sequelae such as limb paralysis should not affect the NIHSS score, and the modified Rankin scale (mRS) score should be ≤1 point.
6. Patient informed consent must be obtained.
7. The criteria for the syndrome of phlegm and blood stasis are as follows: Main syndrome: hemiplegia, mouth and eyes skew, speech retarding or silent, sensation diminished or disappeared; Secondary syndrome: excessive sputum, fat tongue with teeth marks on the side, dark red tongue, sublingual vein blue or tortuous, tongue spots, white or thick greasy fur, pulse slippery.

   -

Exclusion Criteria:

1. subarachnoid hemorrhage, transient ischemic attack, or other intracranial lesions such as intracranial tumor, aneurysm, vascular malformation, cerebral cysticercosis, intracerebral schistosomiasis, encephalitis, meningitis, hydrocephalus, and sequelae of brain trauma; Nonatherosclerotic thrombotic cerebral infarction (e.g., cardiogenic embolism, hypercoagulability disorders, endovascular shedding and arteritis);
2. onset occurring within a range of 30 to 40 days；
3. The patient presents with limb motor dysfunction, emotional disorder, cognitive impairment, or speech impairment resulting from pre-existing conditions (e.g., surgery, trauma, or congenital disability) prior to the onset of cerebrovascular accident.
4. Patients with severe cardiac disease, heart failure, liver or kidney failure, malignant tumors, gastrointestinal bleeding, severe infections, or uncontrolled diabetes are excluded from the study.
5. Individuals currently participating in other clinical trials are not eligible for inclusion.
6. Exclusion criteria include patients with mental illness, multiple body ulcers or joint contractures.
7. Non-compliance with treatment by patients and their families is considered an exclusion criterion.
8. Inability to comprehend the content of informed consent and inability to provide a signature on the informed consent form are also grounds for exclusion.
9. . Pregnant and lactating women are excluded from participation.

   -

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale Score | 0,30days,60days and 90days post-intervention
  Higher scores mean a worse outcome,measured by the overall distribution from 0 (no symptoms) to 6 (death).

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | 0,30days,60days and 90days post-intervention
  Higher scores mean a worse outcome,measured by the overall distribution from 0 (normal) to 42 (severe apoplexy).
Carotid atherosclerotic plaque score | 0 and 90days post-intervention
  Course scoring system for neck carotid atherosclerotic plaque scoring. Higher scores mean a worse outcome,the minimum value is 0 . The plaque score of the carotid artery on each side was calculated by summing up the maximum thickness (mm) of isolated carotid artery plaques, and the total plaque score of each patient was obtained by adding up the plaque scores from both sides.

OTHER OUTCOMES:
Laboratory indicator | 0 and 90days post-intervention
  ① Vascular inflammatory mediators: IL-6, IL-10, and TNF-α in the serum and cell supernatant of each group will be quantified using ELISA.
  ② Reprogramming of lipid metabolism: qRT-PCR will be used to detect metabolic enzymes and transcription factors, including HK,LDH, uPFK-2,PKM,PDK, G6PD, CPT1, ATGL, and HSL.
  ③ Blood lipid: LDL-C,TC, HDL-C and TG.
Score of symptoms and signs in traditional Chinese medicine | 0,30days,60days and 90days post-intervention
  Recovery is defined as a curative effect index ≥90% after treatment; Obvious effect referred to a syndrome efficacy index ≥70% and <90% after treatment; Progress indicated a syndrome efficacy index ≥30% and <70% after treatment; Ineffective denoted a syndrome efficacy index <30% after treatment.
biological indicator | 0,30days,60days and 90days post-intervention
  ① Demographic characteristics: gender, age, educational attainment, stature, body mass index (BMI), occupational status (at baseline).
  ② Fundamental physiological indicators: body temperature, cardiac rhythm, respiration rate, arterial pressure, and glycemic level.
  ③ Previous medical history: the presence of blood pressure, blood glucose, and blood lipid abnormalities, as well as a family history of related diseases.

IPD SHARING:
Plan to Share IPD: Undecided